CLINICAL TRIAL: NCT05679388
Title: A Phase Ib Study of Extending Relugolix Dosing Intervals Through Addition of the CYP3A4 and Pg-P Inhibitor Itraconazole or Ritonavir in Prostate Cancer Patients
Brief Title: A Study of Extending Relugolix Dosing Intervals Through Addition of Itraconazole or Ritonavir in Prostate Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by the PI
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB22-1150
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic; Prostate Adenocarcinoma
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix; Ritonavir; Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Study Group 1 (Experimental): All study participants will receive a starting dose of relugolix (360 mg in the form of three 120 mg tablets) on Day 1 of the 29-day drug administration period. After Day 1, you will receive relugolix on its own or relugolix combined with another medication called itraconazole or ritonavir. The combination of medications you receive, the dosage for each medication, and when you take each medication will be based on the study group you are enrolled in.
  Study Group 1 will receive:
  * Relugolix (360 mg) on Day 1
  * Relugolix (120 mg) on Days 2-7
  Interventions: Drug: Relugolix Pill
- Study Group 2a (Experimental): All study participants will receive a starting dose of relugolix (360 mg in the form of three 120 mg tablets) on Day 1 of the 29-day drug administration period. After Day 1, you will receive relugolix on its own or relugolix combined with another medication called itraconazole or ritonavir. The combination of medications you receive, the dosage for each medication, and when you take each medication will be based on the study group you are enrolled in.
  Study Group 2a will receive:
  * Relugolix (360 mg) on Day 1
  * Relugolix (120 mg) on Days 2-7
  * Itraconazole (200 mg) on Days 1-14
  Interventions: Drug: Relugolix Pill; Drug: Itraconazole
- Study Group 2b (Experimental): All study participants will receive a starting dose of relugolix (360 mg in the form of three 120 mg tablets) on Day 1 of the 29-day drug administration period. After Day 1, you will receive relugolix on its own or relugolix combined with another medication called itraconazole or ritonavir. The combination of medications you receive, the dosage for each medication, and when you take each medication will be based on the study group you are enrolled in.
  Study Group 2b will receive:
  * Relugolix (360 mg) on Day 1
  * Relugolix (120 mg) on Days 2-7
  * Ritonavir (100 mg tablets taken by mouth) on Days 1-14
  Interventions: Drug: Relugolix Pill; Drug: Ritonavir
- Study Group 3a (Experimental): All study participants will receive a starting dose of relugolix (360 mg in the form of three 120 mg tablets) on Day 1 of the 29-day drug administration period. After Day 1, you will receive relugolix on its own or relugolix combined with another medication called itraconazole or ritonavir. The combination of medications you receive, the dosage for each medication, and when you take each medication will be based on the study group you are enrolled in.
  Study Group 3a will receive:
  * Relugolix (360 mg) on Day 1
  * Relugolix (120 mg) on Days 2-4
  * Itraconazole (200 mg tablets taken by mouth) on Days 1-14
  Interventions: Drug: Relugolix Pill; Drug: Itraconazole
- Study Group 3b (Experimental): All study participants will receive a starting dose of relugolix (360 mg in the form of three 120 mg tablets) on Day 1 of the 29-day drug administration period. After Day 1, you will receive relugolix on its own or relugolix combined with another medication called itraconazole or ritonavir. The combination of medications you receive, the dosage for each medication, and when you take each medication will be based on the study group you are enrolled in.
  Study Group 3b will receive:
  * Relugolix (360 mg) on Day 1
  * Relugolix (120 mg) on Days 2-4
  * Ritonavir (100 mg) on Days 1-14
  Interventions: Drug: Relugolix Pill; Drug: Ritonavir

INTERVENTIONS:
Drug: Relugolix Pill — A medication used to treat prostate cancer. Relugolix comes as a tablet to take by mouth. It is usually taken with or without food once daily.
Drug: Ritonavir — HIV antiviral It can treat HIV infection, which causes AIDS. It does not cure HIV or AIDS, but combinations of drugs may slow the progress of the disease and prolong life.
  Arms: Study Group 2b; Study Group 3b
Drug: Itraconazole — A drug used to treat fungal infections.
  Other Names: Sporanox
  Arms: Study Group 2a; Study Group 3a

SUMMARY:
Researchers leading this study hope to learn about the safety of combining the study drug relugolix with another study drug called itraconazole or ritonavir in prostate cancer. This study is for individuals who have advanced prostate cancer and plans to have medical castration (the use of medications or chemicals to lower hormone production in the testicles). Your participation in this research will last up to 1 month.

The purpose of this research is to gather information on the safety and effectiveness of relugolix in combination with ritonavir or itraconazole. The goal of this research is to find out if combining two medications (relugolix and itraconazole or relugolix and ritonavir) could possibly lead to using less relugolix, which is an expensive drug.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed prostate cancer with plans to start medical castration therapy.
* Age 18 or older. Because no dosing or adverse event data are currently available on the use of relugolix in combination with itraconazole or ritonavir in patients <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group performance status ≤2 (Karnofsky ≥60%)
* Participants must satisfy the following laboratory criteria:
* Testosterone > 200 ng/dl
* QTc within normal limits
* Aspartate Transferase (AST)/alanine transaminase (ALT) < 3x upper limit of normal
* Ability to take oral medication and be willing to adhere to the medication regimen.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Need for combination systemic therapy for prostate cancer including docetaxel and/or second-generation androgen receptor pathway targeted agents (i.e. abiraterone, enzalutamide, apalutamide, darolutamide, etc).
* Concurrent therapy with strong interacting drugs with CYP3A4 and P-gp (See Appendix list of strong inhibitors or inducers) due to concerning possible drug-drug interactions with itraconazole, ritonavir and relugolix. Potential drug-drug interactions will also be reviewed by study investigators prior to enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to relugolix, itraconazole or ritonavir.
* Patients receiving treatment with another investigational drug or other intervention within 3 expected half-lives of the agent.
* Serious or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* New York Heart Association Class III of IV congestive heart failure
* Known gastrointestinal malabsorption.
* Active psychiatric illness/social situations that would limit compliance with protocol requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants with prostate cancer.
Enrollment: 60 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Testosterone Suppression of Participants as Assessed by Testosterone Levels | 1 month post start of treatment
  To determine whether the addition of itraconazole and ritonavir to relugolix sustains testosterone suppression as assessed by participant testosterone levels.

SECONDARY OUTCOMES:
Decrease in Relugolix Levels | 1 month post start of treatment
  To evaluate whether itraconazole or ritonavir significantly decreases relugolix clearance in participants with prostate cancer as assessed by relugolix serum levels on days 8 and 15.
Reduction in Prostate-Specific Antigens Levels of Participants After Study Treatment | 1 month post start of treatment
  To evaluate the efficacy of itraconazole or ritonavir combined with relugolix in patients with prostate cancer as assessed by a reduction in Prostate-Specific Antigen (PSA) levels of patients after study treatment.
Rate of Reported Adverse Events Among Participants | 1 month post start of treatment
  To evaluate the safety of itraconazole or ritonavir combined with longer interval relugolix dosing regimens in patients with prostate cancer as assessed by the rate of reported adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) V5.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States